CLINICAL TRIAL: NCT07328438
Title: Diagnosis Disclosure Support Intervention Program for Caregivers of Children With ASD
Brief Title: Diagnosis Disclosure Support for Caregivers of Children With Autism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, So Hyun Kim, Associate Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2025-0578-01; 00209635 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized Waitlist Control Group Design
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Caregivers will participate in an online diagnosis disclosure support intervention delivered via telehealth over five weekly 60-minute group sessions. This program is designed to support caregivers' decision-making and communication regarding disclosure of an ASD diagnosis to their child, including key considerations for disclosure and the development of an individualized narrative to explain the diagnosis. Sessions will include psychoeducation and interactive activities to promote engagement and skill practice.
  Interventions: Behavioral: SHARE : Supporting Honest Autism Recognition and Education
- Waitlist Control Group (Active Comparator): A one-session, group-based psychoeducational seminar delivered via telehealth will be provided to the control group. This abbreviated session will provide a condensed overview of the SHARE program, and caregivers will receive the complete SHARE program materials.
  Interventions: Behavioral: One-session seminar

INTERVENTIONS:
Behavioral: SHARE : Supporting Honest Autism Recognition and Education — Our intervention will consist of a five-week, telehealth-based group intervention (60 minutes per week) to support caregivers of children with ASD (7- to 12-year-olds) regarding diagnosis disclosure. This program provides guidance on the rationale for disclosure, strategies for initiating conversations, and the understanding that disclosure is a gradual, lifelong journey. In addition, the program helps caregivers customize disclosure based on their child's development and emotional readiness. The curriculum moves beyond didactic instruction by combining psychoeducation with experiential, participant-centered activities to support practice and application.
  Arms: Intervention Group
Behavioral: One-session seminar — The control group will receive a 60-minute telehealth seminar providing a condensed overview of the SHARE program and the complete set of SHARE program materials.
  Arms: Waitlist Control Group

SUMMARY:
The purpose of this randomized controlled pilot study is to develop and evaluate an online diagnosis disclosure support intervention for caregivers of 7- to 12-year-old children with autism spectrum disorder (ASD) in South Korea. This intervention is designed to support caregivers who are contemplating, preparing for, or carrying out disclosure of their child's ASD diagnosis to the child. This study has three primary aims: (1) to evaluate the acceptability and feasibility of the intervention; (2) to examine clinically meaningful effects of the intervention on caregivers' psychological well-being and psychosocial adjustment (e.g., emotion regulation, loneliness/social isolation, and adaptation to life transitions), parenting competence and attitudes (e.g., parenting self-efficacy, parenting role satisfaction, and parenting stress), and autism-related knowledge and social perceptions (e.g., autism knowledge and perceived autism-related stigma); and (3) to assess whether the effects of the intervention are maintained one month after program completion.

DETAILED DESCRIPTION:
As school-aged children with autism spectrum disorder begin to recognize differences between themselves and their neurotypical peers, they develop questions regarding their identity and belonging. During this critical developmental period, receiving a clear and supportive explanation of their diagnosis can promote self-understanding, encourage self-advocacy, and enhance psychosocial adjustment. However, caregivers often face significant barriers to disclosing the diagnosis, stemming from fear of stigma, uncertainty about appropriate timing and language, and concerns about causing emotional distress. As a result, caregivers may delay or avoid disclosure, despite potential benefits for the child. Therefore, developing evidence-based interventions to support caregivers in diagnosis disclosure is significant, yet few studies offer guidance for caregivers, leaving disclosure decisions and processes largely to individual families.

The purpose of this randomized controlled pilot study is to develop and evaluate an online diagnosis disclosure support intervention for caregivers of 7- to 12-year-old children with ASD in South Korea, a developmental period when children go through increasing cognitive, social, and identity-related challenges. This study pursues three objectives: (1) to evaluate the acceptability and feasibility of the diagnosis disclosure support intervention; (2) to examine clinically meaningful effects on caregiver's outcomes across domains such as psychological well-being and psychosocial adjustment, parenting competence and attitudes, and autism-related knowledge and social perceptions; and (3) to assess the sustainability of these effects through a one-month follow-up after program completion.

40 caregivers of children with ASD enrolled in mainstream schools (grades 2-6) in South Korea will be recruited and randomly assigned to either an intervention group (n=20) or a waitlist control group (n=20). The intervention group will participate in a five-week, online group-based diagnosis disclosure support program consisting of weekly 60-minute sessions, which will be recorded for fidelity monitoring. The waitlist control group will receive an abbreviated one-session online seminar and program materials upon completion of the final follow-up assessment. Both groups will complete online self-report measures at three timepoints: baseline (T1), immediately following the intervention group's program completion (T2), and at a one-month follow-up (T3). This study holds the potential to improve caregivers' well-being and support healthy family communication by providing evidence-based guidance to facilitate developmentally appropriate disclosure for children with ASD in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children aged 7-12 (Grades 2-6) attending mainstream schools in South Korea
* Caregivers of children with previous medical diagnosis of ASD
* Caregivers with no prior experience of participation in diagnosis disclosure support programs
* Caregivers in agreement with the need for a ASD diagnosis disclosure support intervention program, with commitment to continuous and sincere participation

Exclusion Criteria:

* Caregivers of children with significant intellectual disability
* Caregivers of children with significant language delay

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Parental Autism Disclosure Scale (PADS) | baseline, immediately after the intervention, 1-month follow-up
  The Parental Autism Disclosure Scale (PADS) is a self-report instrument developed in this study to measure the extent to which caregivers of autistic children have considered and prepared for disclosing the diagnosis to their child. The scale consists of 26 items rated on a 5-point Likert scale ranging from "strongly disagree" (0) to "strongly agree" (4), with reverse-scored items included. Higher total scores indicate greater consideration of and preparedness for disclosing the diagnosis to the child, with total scores ranging from 0 to 104.
Decisional Conflict Scale (DCS) | baseline, immediately after the intervention, 1-month follow-up
  The Decisional Conflict Scale (DCS) will be used to assess decision-making conflict regarding diagnosis disclosure among caregivers of children with autism. Items are rated on a 5-point Likert scale ranging from "strongly agree" (0) to "strongly disagree" (4). Total scores and subscale scores are converted to a 0-100 scale, with higher scores indicating greater decisional conflict.
Diagnosis Disclosure Support Intervention Program Acceptability Survey | immediately after the intervention
  This will be used to assess whether the intervention program was satisfying and comprehensible to caregivers. Caregivers will respond to approximately 10 items using a Likert-type scale. The survey will include items such as "The program fits the goals of the intervention" and "The skills taught in the program are relevant to my needs."
Diagnosis Disclosure Support Intervention Program Feasibility Survey | immediately after the intervention
  This will be used to assess whether the intervention program was feasible for the caregivers. Caregivers will respond to approximately 10 items using a Likert-type scale. The survey will include items related to the practicality of the program such as 'Using Zoom for the sessions was easy for me.' and 'The length of each session was manageable.'
Participation Survey | during each of the five sessions (weeks 1 to 5) in intervention program
  A form will be used to record the attendance of the caregivers as a measure of their participation in the intervention program.
Intervention Fidelity Checklist | every 3 months from the start of the intervention for each therapist
  This will be used to assess whether core elements in each session were delivered to caregivers. Interventionists will record the checklist for each session.

SECONDARY OUTCOMES:
Korean Version of Internalized Stigma of Mental Illness Scale (K-ISMI) | baseline, immediately after the intervention, 1-month follow-up
  The Korean Version of the Internalized Stigma of Mental Illness Scale (K-ISMI) will be used to measure the level of internalized stigma experienced by caregivers and to assess the impact of stigma on family stress and adaptation. Items are rated on a 4-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (4), with reverse-scored items included. Total scores range from 29 to 116, with higher scores indicating a higher level of internalized stigma related to having a child with autism.
Life Transition Scale for Parents of Children with Autism (LTS) | baseline, immediately after the intervention, 1-month follow-up
  The Life Transition Scale for Parents of Children with Autism (LTS) will be used to assess the emotional responses and psychological adaptation of caregivers of autistic children during the process of recognizing and accepting their child's diagnosis. Items are rated on a 4-point Likert scale ranging from "never" (1) to "often" (4), with reverse-scored items included. Evaluation of the transition process is conducted by calculating the mean score for each stage, obtained by dividing the sum of item scores within each stage by the number of items; higher or lower mean scores are then compared across stages.
Emotion Regulation Questionnaire (ERQ) | baseline, immediately after the intervention, 1-month follow-up
  The Emotion Regulation Questionnaire (ERQ) will be used to assess how caregivers experience and regulate their emotions in their daily lives. Items are rated on a 7-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (7). Higher scores indicate greater use of the corresponding emotion regulation strategy.
Autism Stigma and Knowledge Questionnaire (ASK-Q-2) | baseline, immediately after the intervention, 1-month follow-up
  The Autism Stigma and Knowledge Questionnaire (ASK-Q-2) will be used to assess caregivers' knowledge of and stigma toward autism. Items are scored dichotomously (agree = 1, disagree = 0).
Parenting Sense of Competence (PSOC) | baseline, immediately after the intervention, 1-month follow-up
  The Parenting Sense of Competence (PSOC) scale is a parent self-report measure used to assess parenting satisfaction and efficacy. Items are rated on a 6-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (6), with reverse-scored items included. Higher total scores indicate greater parental efficacy. Scores of 58 or below are interpreted as low, scores between 58 and 74 as average, and scores of 75 or above as high.
Parent Satisfaction Scale (PSS) | baseline, immediately after the intervention, 1-month follow-up
  The Parent Satisfaction Scale (PSS) is an instrument that assesses caregivers' subjective evaluation of their performance in the parenting role, as well as the positive and negative emotions arising from their parenting experiences. Items are rated on a 4-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (4), with reverse-scored items included. Higher total scores indicate greater satisfaction with the parenting role.
Korean Parenting Stress Index Fourth Edition Short Form (K-PSI-4-SF) | baseline, immediately after the intervention, 1-month follow-up
  The Korean Parenting Stress Index-Fourth Edition Short Form (K-PSI-4-SF) is a parent self-report measure used to assess parenting stressors and overall levels of parenting stress. Items are rated on a 5-point Likert scale with varying anchor statements (e.g., from "strongly disagree" (1) to "strongly agree" (5); from "definitely not adequate as a parent" (1) to "a very good parent" (5); and from "much easier than expected" (1) to "much more difficult than expected" (5)). Total scores range from 36 to 180, with higher total scores indicating greater levels of stress experienced in parenting.
UCLA Loneliness Scale-8 (ULS-8) | baseline, immediately after the intervention, 1-month follow-up
  The UCLA Loneliness Scale-8 (ULS-8) is a self-report measure that assesses the degree and frequency of perceived loneliness and will be used to measure loneliness as a state of extreme distress resulting from relational deficiency. Items are rated on a 4-point Likert scale ranging from "strongly disagree" (1) to "always" (4), with reverse-scored items included. Total scores range from 8 to 32, with higher total scores indicating higher levels of perceived loneliness.
Loneliness and Social Isolation Scale (LSIS) | baseline, immediately after the intervention, 1-month follow-up
  The Loneliness and Social Isolation Scale (LSIS) is an instrument designed to estimate the complex construct of social isolation by incorporating both objectively measurable aspects of social networks and individuals' subjective perceptions of social support and loneliness. Items 1 and 2 are rated on a scale ranging from "rarely true" (0) to "very true" (3). Items 3 and 4 are reverse-scored, ranging from "rarely true" (3) to "very true" (0). Item 5 assesses the number of social contacts, scored from "0 persons" (3) to "7 or more persons" (0), and Item 6 assesses time spent in social interaction, scored from "not at all" (3) to "1 hour or more" (0). A total score of 3 or higher on Items 1 and 2 indicates a high risk of loneliness. A total score of 4 or higher on Items 3 and 4, together with a total score of 4 or higher on Items 5 and 6, indicates a high risk of social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: So Hyun Kim, Ph.D., Principal Investigator — Korea University; Kyoung Hong, Ph.D., Study Director — Korea University